CLINICAL TRIAL: NCT05883527
Title: Partnership in Safeguarding People With Dementia From Primary and Social Care Perspectives
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Reena Lasrado, Principal Investigator, University of Manchester
Other Study IDs: IRAS ID: 319897
Record Dates: First submitted 2023-05-10; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Dementia; Abuse Client; Neglect; Care, Malnutrition
Keywords: Safeguarding; Abuse; Neglect; Dementia; Health and care professionals; Social care; Section 42
MeSH Terms: conditions — Dementia; Malnutrition | interventions — Caregivers

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Health and Care Professionals: GP's, nurses, social workers, mental health professionals, support workers, Independent mental capacity advocates (IMCA), and other HCP's working in GP surgeries and integrated social care hubs. Safeguarding leads in GP surgeries, social care organisations and other relevant organisations. Professionals from third-sector organisations who have previous experience of safeguarding.
  Interventions: Other: Not applicable as not an intervention - HCP's
- People Living with Dementia: Who have been involved in the safeguarding process and have capacity to consent.
  Interventions: Other: Not applicable as not an intervention - PLwD and family/carers
- Paid carers of people living with dementia: Who have been involved in the safeguarding process.
  Interventions: Other: Not applicable as not an intervention - PLwD and family/carers
- Family members of people living with dementia: Who have been involved in the safeguarding process.
  Interventions: Other: Not applicable as not an intervention - PLwD and family/carers

INTERVENTIONS:
Other: Not applicable as not an intervention - PLwD and family/carers — Exploring the safeguarding process through interviews.
  Groups: Family members of people living with dementia; Paid carers of people living with dementia; People Living with Dementia
Other: Not applicable as not an intervention - HCP's — Exploring the safeguarding process through interviews and a focus group.
  Groups: Health and Care Professionals

SUMMARY:
"Adult safeguarding is everyone's responsibility". The Care Act 2014 makes safeguarding a legal duty. It provides local authorities and other agencies in England with a responsibility to protect adults with care and support needs from abuse and neglect. This is done most effectively when all relevant agencies work together. This is particularly important for people living with dementia, as they are at higher risk of abuse or neglect. Such abuse is most common in their own homes and care settings. Primary and social care professionals are likely to have regular contacts with older people, hence have opportunities for early identification and prevention of abuse. However, little is known about how primary care practitioners work in partnership with social care and other agencies to investigate and manage abuse.

Aims:

This project will outline how health professionals in primary care settings understand and respond to abuse and what their understandings of safeguarding law and policy are. It will also identify how social services departments assess and manage referrals relating to people living with dementia in primary care settings. Furthermore, the study will analyse the experiences of people with dementia and families who are at the centre of safeguarding

Methods:

This study has three phases. In phase 1, the investigators will synthesise current research and practice evidence to develop a theory of safeguarding conceptualisation and process. In phase 2, the investigators will analyse national statistics on safeguarding (NHS digital dataset), ageing and dementia data (English Longitudinal Study of Ageing) to understand patterns of reporting and how they vary across location, gender, ethnicity and time period. In phase 3, the investigators will interview GPs, social workers, safeguarding leads, independent advocates, people with dementia, family members, support workers, carers and other professionals who make or receive referrals via primary care. As part of phase 3 group discussions will also be conducted, in which professionals will come together to share their experiences, and will identify approaches for preventing abuse and collaboration amongst relevant agencies. Phase 3 will inform the development of complex case studies, drawing on data from phases 1 and 2.

Impact:

This study will help develop practice guidance for professionals, to aid multi-agency collaboration in safeguarding cases specific to dementia. This will be developed in consultation with the PPIE (Patient and Public Involvement and Engagement) members and practitioners. Videos will also be produced and plain English versions of case studies of complex safeguarding scenarios and strategies in consultation with safeguarding leads, law experts, training providers and other key stakeholders. Experts by experience (working with, caring for or living with dementia), will be able to guide the team with cultural nuances and appropriateness to ensure that the material developed is sensitive to all populations. An info graph/pictograph displaying signs of abuse, staying safe and what to do, aimed at people with dementia and family will be compiled. The investigators will liaise with national safeguarding leads so that this information can be displayed in GP clinics. Furthermore, the investigators will contact social responsibility personnel for supermarkets and discuss the potentials of wider circulation for displaying this information in stores.

ELIGIBILITY:
Inclusion Criteria:

* Health and social care professionals:

  * GPs, Nurses, social workers, mental health professionals, support workers, IMCA (independent mental capacity advocates) and other health care professionals in GP surgeries and integrated social care hubs with experience in facilitating safeguarding.
  * Safeguarding lead in GP surgeries, social care organisations and other organisations (advocacy agencies).
  * Professionals from third-sector organisations who have previously raised safeguarding concerns regarding adults living with Dementia

Service users and carers/family:

* People with dementia who have been involved in the safeguarding process, with mental capacity to consent.
* Family members of people with dementia who have been previously involved in the safeguarding process
* Individuals who were involved in a safeguarding inquiry in the past, which is NOT ongoing at the time of interview.

Exclusion Criteria:

* Health and social care professionals at GP practices, social care organisations and third sector organisations without experiences of safeguarding older adults and unwilling to participate in the study.

  * People with dementia who lack capacity to consent.
  * Individuals involved in an active and ongoing safeguarding inquiry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Tentatively this study will aim to recruit 20-30 health and social care professionals (interviews-20, focus groups-10) making referrals via GP's who have experiences of safeguarding in the context of dementia. This study also aims to recruit between 15-20 people with dementia and carers/family members involved in safeguarding, who will be accessed via primary and social care practitioners.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Trends in reporting of routinely collected safeguarding datasets - NHS digital | September 2022 - March 2024
  Number of reports of safeguarding concerns and section 42 enquiries in England. Type of risks, source of risks, location, age, gender, ethnicity, health condition.
Trends in reporting of routinely collected safeguarding datasets - ELSA data | data years: 2002-2017
  The prevalence of dementia across England, number of older people with dementia in receipt of care and who gave the care in each local authority in England.
Quality Outcomes Framework (QOF) Recorded Dementia Diagnoses | data years: 2021-2022
  Rate of dementia diagnosis in each local authority district in England and demographic characteristics of those with dementia diagnosis in each NHS CCG in England.

OTHER OUTCOMES:
Contexts, Mechanisms and Outcomes (CMO's) from the Rapid Realist Literature Review | September 2022 - March 2024
  The rapid realist review will investigate how health & social care professionals conceptualise and respond to risks of abuse and neglect involving people with dementia in England, UK. The review will be informed by Rameses guidelines and aims to develop initial programme theories.
Interpretative Phenomenological Analysis (IPA) of Interviews | September 2022 - March 2024
  IPA of interview transcripts will lead to an in-depth understanding of the lived experiences of safeguarding from the perspective of health and social care professionals, people living with dementia, family caregivers and other relevant professionals.
Interpretative Phenomenological analysis (IPA) of Focus Group - with health and care professionals | September 2022 - March 2024
  Lived experiences of safeguarding from the perspective of various professionals, including what worked, what did not work, understanding of legal thresholds, strategies for prevention and collaboration across agencies.

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - CRN, Leeds
  - Leeds Local Authority, Leeds
  - CRN, Manchester
  - Greater Manchester Local Authority, Manchester
  - CRN, Southport

IPD SHARING:
Plan to Share IPD: Undecided